CLINICAL TRIAL: NCT07002749
Title: ROLE OF PROPHYLACTIC TRANEXAMIC ACID IN PREVENTION OF POST-PARTUM HEMORRHAGE IN ELLSCS
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Patel Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, NIMRA ABID CHAUHAN, RESIDENT OBGYN, Patel Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PH/IRB/2025/002
Record Dates: First submitted 2025-05-18; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Active Comparator): tranexamic acid
  Interventions: Drug: Tranexamic Acid (TXA)
- B (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — I would like to see the effect of prophylactic tranexamic acid in women undergoing ELLSCS in preventing PPH in my setup.
  Arms: A
Device: Placebo — one group will get placebo
  Arms: B

SUMMARY:
IN THIS STUDY WOMEN UNDER GOING ELLSCS WOULD BE DIVIDED INTO TWO GROUPS , ONE GROUP WOULD BE GIVEN TRANEXAMIC ACID WHILE THE OTHER WOULD BE GETTING PLACEBO PROPHYLACTICALLY TO SEE THE EFFECT OF TRANEXAMIC ACID IN PREVENTING PPH.

THIS IS A RANDOMIZED CONTROLLED TRIAL. THE SAMPLING TECHNIQUE WOULD BE NON-PROBABILITY TECHNIQUE RANDOMIZATION WOULD BE DONE VIA BALLOTING METHOD.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with singleton pregnancy and low risk for PPH admitted for ELLSCS

Exclusion Criteria:

Women with medical disorder or complex pregnancy.

* Women with history of PPH.
* Women with bleeding disorder.
* Abnormal placentation (MAP, placenta previa)
* Multiple pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 104 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
prophylactic tranexamic acid in prevention of post-partum haemorrhage in ELLSCS | 6 months from the time of approval from CPSP till the completion of data collection
  In this study, the role of tranexamic acid is being observed in preventing PPH in women undergoing ELLSCS by dividing women into two groups and giving one group placebo while the other would receive tranexamic acid.
  Two boxes, A and B, each containing 52 vials of the same size and color; one would contain the drug, i.e: TXA 1000 mg in 10 ml , while the other would contain a placebo in 10 ml vial, provided by a company; these would be revealed at the end of the study. A jar containing 104 chits, 52 of which would have the letter A written on them and the other 52 would have the letter B, would be kept in GYNAE OT. Prior to ELLSCS, a chit would be selected from the jar, and the patient would be given the drug according to the chit. It's a triple-blinded study; the patient, doctor, surgeon, and data analyst all will be blinded.

CONTACTS AND LOCATIONS:
Locations (1):
- Patel Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37292548/